CLINICAL TRIAL: NCT01470898
Title: Effect of Bispectral Index (BIS) Monitoring on Faster Recovery Time and Analgesic Consumption in Abdominal Surgery Patients
Brief Title: Bispectral Index (BIS) Monitoring in Abdominal Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Jasminka Persec, MD, PhD, MD PhD, University Hospital Dubrava
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 12377KBD
Record Dates: First submitted 2011-11-07; First posted 2011-11-11 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2011-11

CONDITIONS: Anesthesia
Keywords: bispectral index monitoring; extubation; analgesia; abdominal surgery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- anesthesia monitoring (Experimental): Bispectral Index Monitoring (BIS) has been proven to be effective in preventing awareness. Optimizing anesthesia level using BIS monitoring, neither to light nor to deep will probably help to shorten recovery time and reduce drug consumption. A BIS sensor was applied to patient's forehead before induction of anesthesia and connected to A-2000 BIS monitor (Aspect Medical Systems, Newton, MA, USA). It records the electroencephalogram from 4 electrodes and after processing it with mathematic algorithms it generates a number from 0 to 100. When the BIS value is lower than 40, the patient is in deep anesthesia state, when the value is over 80, the patient is under light sedation.
  Interventions: Device: bispectral index monitoring
- no bispectral index monitoring (Experimental): At the induction of anesthesia, and every 15 minutes during operation following parameters were recorded: heart rate (HR), systolic blood pressure (BP), end-tidal CO2 (etCO2) and BIS level. Also, operation time and extubation time were recorded. Finally, all patients were visited on the first postoperative day and interviewed about intraoperative recall.
  Interventions: Device: bispectral index monitoring

INTERVENTIONS:
Device: bispectral index monitoring — A BIS sensor was applied to patient's forehead before induction of anesthesia and connected to A-2000 BIS monitor (Aspect Medical Systems, Newton, MA, USA). It records the electroencephalogram from 4 electrodes and after processing it with mathematic algorithms it generates a number from 0 to 100. When the BIS value is lower than 40, the patient is in deep anesthesia state, when the value is over 80, the patient is under light sedation.At the induction of anesthesia, and every 15 minutes during operation following parameters were recorded: heart rate (HR), systolic blood pressure (BP), end-tidal CO2 (etCO2) and BIS level. Also, operation time and extubation time were recorded. Finally, all patients were visited on the first postoperative day and interviewed about intraoperative recall.

SUMMARY:
Bispectral Index Monitoring (BIS) has been proven to be effective in preventing awareness. Optimizing anesthesia level using BIS monitoring, neither to light nor to deep will probably help to shorten recovery time and reduce drug consumption. The aim of the study was to investigate the effect of BIS monitoring on extubation and recovery time, and intraoperative anesthesia consumption.

DETAILED DESCRIPTION:
Patients undergoing major abdominal surgery under general anesthesia in University Hospital Dubrava, were eligible if there were aged 18 years or older, and ASA (American Society of Anesthesiologists) physical status II or III. Study included 40 patients enroled in the six months period (between February 2011. and July 2011.). Exclusion criteria were memory impairment, psychosis, known or suspected electroencephalograph abnormality (eg, epilepsy, previous brain operation), chronic use of psychoactive medication, and operation time exceeding six hours.

The protocol was approved by Institutional Ethics Committee of University Hospital Dubrava. All participating elective surgical patients were given brief description of the trial, and gave written informed consent before enrolment.

According to a computer generated randomisation list, patients were randomly assigned to receive BIS-guided anesthesia (group 1) or routine anesthesia care as a non BIS-guided group (group 2). The non BIS-guided group was studied while the BIS monitor was attached to patient, but the screen was blinded to the anesthesiologist in charge. All values were recorded by the younger anesthesiologist, who was not involved in the anesthesia maintenance. All other aspects of perioperative treatment were similar, including choice of anesthetic agents and monitoring.

The operation was performed under general anesthesia using midazolam (0.15 mg/kg), fentanyl (2 µg/kg) and pancuronium (0.1 mg/kg) to facilitate endotracheal intubation, and 1.5-2.5 MAC of sevoflurane, nitrous oxide 50% in oxygen, boluses of fentanyl and pancuronium for maintenance. Intraoperatively, after induction doses of fentanyl, anesthesia was mainly balanced with sevoflurane. Electrocardiography (EKG), invasive blood pressure (IBP), peripheral oxygen saturation (SpO2), and end-tidal CO2 (etCO2) were monitored.

A BIS sensor was applied to patient's forehead before induction of anesthesia and connected to A-2000 BIS monitor (Aspect Medical Systems, Newton, MA, USA). It records the electroencephalogram from 4 electrodes and after processing it with mathematic algorithms it generates a number from 0 to 100. When the BIS value is lower than 40, the patient is in deep anesthesia state, when the value is over 80, the patient is under light sedation [3].

After the surgery and recovery from anesthesia, patients were transferred to intensive care unit for continuous monitoring of vital functions and homeostasis.

At the induction of anesthesia, and every 15 minutes during operation, BIS levels were recorded. Also, at the end of the operation, extubation time and analgesics consumption were recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing major abdominal surgery under general anesthesia in University Hospital Dubrava, were eligible if there were aged 18 years or older
* ASA (American Society of Anesthesiologists) physical status II or III.

Exclusion Criteria:

* memory impairment,
* psychosis,
* known or suspected electroencephalograph abnormality (eg, epilepsy, previous brain operation),
* chronic use of psychoactive medication,
* operation time exceeding six hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-07 (Actual); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Bispectral index (BIS) monitoring in abdominal surgery patients | six months
  At the induction of anesthesia, and every 15 minutes during operation BIS levels were recorded.

SECONDARY OUTCOMES:
Effect of bispectral index (BIS) monitoring on faster recovery time in abdominal surgery patients | six months
  At the end of operation, time to extubation were measured.

CONTACTS AND LOCATIONS:
Overall Officials: Jasminka Persec, MD PhD, Principal Investigator — Anesthesiology, reanimatology and intensive care medicine Clinic, University Hospital Dubrava, Zagreb, Croatia; Zoran Persec, MD PhD, Study Chair — Department of urology, University Hospital Dubrava, Zagreb, Croatia; Ino Husedzinovic, Professor, Study Director — Head of Anesthesiology, reanimatology and intensive care medicine Clinic, University Hospital Dubrava, Zagreb, Croatia
Locations (1):
- University Hospital Dubrava, Zagreb, Croatia

REFERENCES:
- [Derived] Persec J, Persec Z, Kopljar M, Sojcic N, Husedzinovic I. Effect of bispectral index monitoring on extubation time and analgesic consumption in abdominal surgery: a randomised clinical trial. Swiss Med Wkly. 2012 Oct 9;142:w13689. doi: 10.4414/smw.2012.13689. eCollection 2012. PMID 23135976